CLINICAL TRIAL: NCT00154687
Title: A Phase II Study of Weekly Paclitaxel, Cisplatin and 24-Hour Infusion of High-Dose 5-Fluorouracil and Leucovorin(Weekly TP-HDFL) in the Treatment of Advanced Transitional Cell Carcinoma(TCC)
Brief Title: Weekly TP-HDFL in the Treatment of Advanced TCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 159I3
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2005-07

CONDITIONS: Transitional Cell Carcinoma
Keywords: Combination, Chemotherapy,transitional cell carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Paclitaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Paclitaxel, Cisplatin, 5-Fluorouracil

INTERVENTIONS:
Drug: Paclitaxel, Cisplatin, 5-Fluorouracil

SUMMARY:
The purpose of this study is to evaluate the efficacy of Weekly TP-HDFL in advanced transitional cell carcinoma in terms of response rate and overall survival.

DETAILED DESCRIPTION:
Transitional cell carcinoma(TCC)of urothelium,including bladder, ureter, and renal pelvis TCCs, was the most lethal urology malignancy in Taiwan. In 1995, approximately 1,300 new cases of TCC was diagnosed in Taiwan and more than 600 patients died of this disease. Advanced TCC is a moderately chemosensitive disease. A combination of methotrexate, vinblastine, and cisplatin with or without doxorubicin (M-VAC or CMV) has been widely used since 1980s. Despite the response rate was as high as 40-70%, the survival of these patients was only slightly increased from a median of 7 to 9 months for those who were treated with supportive care or cisplatin alone to a median of 12 months by cisplatin-based combination chemotherapy. One of the reasons for the poor treatment results is the inevitable treatment-related toxicities related to conventional systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathology proven TCC Recurrent or metastatic TCC Muscle-invasive TCC
2. Measurable disease
3. Age>18
4. KPS>60﹪
5. Creatinine clearance>35ml/min,
6. AST/ALT < or = 3.5times upper limits of normal reference values
7. Bilirubin< or = 2.0 mg/dl
8. WBC > or = 4,000/mm3, PLT > or = 100,000/mm3
9. Written informed consent

Exclusion Criteria:

1. Previous systemic chemo is not allowed
2. TG <70mg/dl
3. CNS metastasis
4. Life expectancy less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2000-10; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
response rate | 2000~2005

SECONDARY OUTCOMES:
Overall Survival ,Safety | 2000~2005

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Hsu, M.D.,Ph.D., Principal Investigator — Department of Oncology , National Taiwan University Hospital; Ann-Lii Cheng, M.D.,Ph.D, Study Chair — Department of Oncology, National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan